CLINICAL TRIAL: NCT03670212
Title: Neuropharmacological Investigation of Frontostriatal Network Function and Nicotine Seeking Behavior in Current Smokers
Brief Title: Investigation of Nicotine Seeking Behavior in Current Smokers
Acronym: NSS
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Wayne State University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Eric Andrew Woodcock, Doctoral Candidate, Wayne State University
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Basic Science
Other Study IDs: 1501013735; F31DA040369 (NIH)
Record Dates: First submitted 2018-09-09; First posted 2018-09-13 (Actual); Last update posted 2018-09-13 (Actual); Status verified 2018-09

CONDITIONS: Cigarette Smoking
Keywords: cigarette smoking; acute stress; executive function; craving; nicotine seeking; relapse; excitatory neural activity; glutamate; negative affect
MeSH Terms: conditions — Cigarette Smoking; Recurrence | interventions — Yohimbine; Hydrocortisone

STUDY DESIGN:
Intervention Model Description: Double-blind, placebo-controlled, and randomized cross-over study design. Each subject completed both the placebo and acute stress experimental sessions.
Who Masked: Participant, Investigator
Masking Description: Double-blinded study. Subjects, the experimenter, research assistants, and MRI technician did not know if the oral doses were active (acute stress condition) or inert (placebo session).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Placebo (Placebo Comparator): The placebo compound, Lactose Monohydrate Powder, was encapsulated in generic opaque capsules identical to the capsules used in the acute stress session. During the placebo session, two capsules were self-administered (swallowed) by each subject. At 11:45am, subjects self-administered a capsule containing 54mg of lactose. At 12:15pm, subjects self-administered a capsule containing 10mg of lactose.
  Interventions: Drug: Lactose Monohydrate Powder
- Acute Stress (Experimental): During the acute stress experimental session, subjects self-administered two generic opaque capsules. At 11:45am, subjects self-administered a capsule containing 54mg of Yohimbine Hydrochloride powder. At 12:15pm, subjects self-administered a capsule containing 10mg of Hydrocortisone.
  Interventions: Drug: Yohimbine Hydrochloride; Drug: Hydrocortisone

INTERVENTIONS:
Drug: Yohimbine Hydrochloride — 54mg of yohimbine powder was encapsulated in a generic opaque capsule and swallowed with water.
  Other Names: YOH
  Arms: Acute Stress
Drug: Hydrocortisone — 10mg hydrocortisone was encapsulated in a generic opaque capsule and swallowed with water.
  Other Names: HYD
  Arms: Acute Stress
Drug: Lactose Monohydrate Powder — Lactose powder was encapsulated in generic opaque capsules identical to those used during the acute stress session. Lactose doses weighed the same as the acute stress session doses (54mg and 10mg, respectively).
  Other Names: Placebo
  Arms: Placebo

SUMMARY:
In this study, 21 non-treatment-seeking cigarette smokers were recruited to investigate the effects of acute stress on brain function and nicotine seeking/self-administration behavior.

DETAILED DESCRIPTION:
Non-treatment-seeking cigarette smoking individuals were recruited from the Detroit, MI area. Individuals were screened for cardiovascular, neurological, and psychiatric contraindications. 21 healthy smokers completed two oral pre-treatment experimental sessions (on separate non-consecutive days) in randomized order under double-blind conditions: placebo (lactose) and stress (54mg yohimbine and 10mg hydrocortisone). Yohimbine + hydrocortisone elicit a neurochemical and physiological response that mimics a 'natural' stressor. Placebo and stress sessions were identical and started at 11am. Upon arrival, subject sobriety was confirmed with expired breath alcohol measurement (<.02%). At 11:30am, each subject smoked 6 cigarette puffs (preferred brand; provided by study) over 5 minutes to control for recent nicotine exposure. Throughout each experimental session, subjects periodically completed self-reported measures of cigarette craving, nicotine withdrawal symptoms, affect, and anxiety, and vital signs were measured. Subjects self-administered (swallowed) oral doses of yohimbine (or placebo) at 11:45am and hydrocortisone (or placebo) at 12:15pm. At 1pm, subjects completed a 60-min neuroimaging scan which included: 1) T1-weighted structural scan, 2) proton functional magnetic resonance spectroscopy (fMRS) acquisition from the left prefrontal cortex during a letter 2-back working memory paradigm, and 3) functional magnetic resonance imaging (fMRI) acquisition during an N-back paradigm yoked with cigarette cues. At 2:30pm, subjects completed an 11-trial choice progressive ratio task in which they could earn cigarette puffs (preferred brand; provided by study) or money. At 3pm, subjects self-administered earned cigarette puffs (video monitored). Subjects remained on site until 4pm discharge.

ELIGIBILITY:
Inclusion Criteria:

* 1) Aged between 21-35 years old, 2) current smokers (expired breath carbon monoxide > 4ppm, self-reported 10+ cigarettes/day, Fagerstrom test for nicotine dependence score > 3, 3) normal seated and resting vital signs (systolic blood pressure 80-160mmHg, diastolic blood pressure 50-90mmHg, and heart rate 50-90 bpm), and 4) normal or corrected-normal vision.

Exclusion Criteria:

* 1) Abnormal electrocardiogram (reviewed by licensed cardiologist), 2) magnetic resonance imaging contraindications (e.g. metal implants), 3) medical/neurological contraindications (e.g., diabetes or head trauma), 4) pregnancy (urine test; females only), 5) positive urine test result for opioids, cocaine metabolites, benzodiazepines, barbiturates, or amphetamines, 6) psychiatric contraindications (subject met criteria for current Axis 1 disorder [other than nicotine dependence] as indicated by computerized MINI-6 screen), and 7) self-reported marijuana and/or alcohol use on 15+ days in the past month.

Ages: 21 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2016-01-07 (Actual); Primary Completion 2016-10-04 (Actual); Study Completion 2016-10-04 (Actual)

PRIMARY OUTCOMES:
Cigarette puff vs. money choice task | 30 minutes
  Participants could earn (via computer mouse 'clicks') money or cigarette puffs (preferred brand; provided by the study) across 11 independent choice trials. At the start of each trial, subjects selected either money or cigarette puffs on a computer screen. After each selection, subjects could earn one unit of that selection by satisfying the computer 'mouse' click requirement. The click requirement increased with each successive unit earned separately for cigarette puffs and money following a progressive ratio schedule (5, 12, 33, 100, 180, 340, 540, 835, 1220, 1660, and 2275 'mouse' clicks; identical schedule for both options and experimental sessions). Units were $0.25 money and 1 cigarette puff. Earned cigarette puffs were smoked at the end of the task and earned money was applied to the subject's study payment. The task was completed between 2:30pm and 3pm for each session.

SECONDARY OUTCOMES:
Letter 2-back task | 12 minutes
  Participants completed 5 blocks of a letter 2-back working memory task during proton functional magnetic resonance spectroscopy data acquisition from the left dorsolateral prefrontal cortex. The 2-back task consisted of a neurochemistry normalization period (passive viewing of a 3Hz flashing checkerboard; 208s) and alternating periods of passive visual fixation (centered fixation cross; 32s) and letter 2-back (64s; 4s instructions ['2-back'], 20 letters [3s/letter; 500ms on screen; 2500ms blank screen], 6 target letters). Changes in neurochemistry as quantified using LCModel were the primary outcome variable. 2-back response accuracy (% correct) and response latency (ms) were secondary outcomes.
Cigarette-cued letter N-back task | 15 minutes
  Participants completed a neutral image vs. cigarette smoking-related image cued letter N-back task during functional magnetic resonance imaging acquisition. The task consisted of pseudo-randomly ordered blocks of 0-, 1-, and 2-back with either cigarette cues or matched neutral images behind each letter. Two 32s blocks of each task permutation were collected separated by 16s of blank screen (to minimize carry-over effects). Patterns of brain activation throughout the task was the primary outcome measure while N-back response accuracy (% correct) and response latency (ms) were secondary outcomes.

OTHER OUTCOMES:
Minnesota Nicotine Withdrawal Scale | 1 minute; collected five times throughout each experimental session
  Well-validated self-report measure of nicotine withdrawal symptoms was measured (MNWS; Hughes and Hatsukami, 1986). Subjects were asked to rate 15 adjectives describing common nicotine withdrawal symptoms on a 5-point Likert scale reflecting symptom severity during the past 10 minutes from 0='not present' to 4='severe'. Mean scores were calculated across items with higher values (maximum=4) reflecting greater withdrawal symptom severity and lower scores (minimum=0) reflecting less severe withdrawal symptoms.
Brief Questionnaire of Smoking Urges | 1 minute; collected five times throughout each experimental session
  Well-validated self-report measure of subjective cigarette craving was measured (QSU; Cox et al., 2001). The self-report measure consists of 10-items with first-person statements describing one's desire to smoke a cigarette. Items are rated on a 7-point Likert scale: 1='strongly disagree' to 7='strongly agree'. Two sub-scales were considered separately; appetitive vs. relief-motivated craving. Sub-scales were quantified as a sum of items: higher scores reflected greater cigarette craving (both sub-scale scores range=5-35).
State-Trait Anxiety Inventory | 1 minute; collected five times throughout each experimental session
  Well-validated self-report measure of state anxiety symptoms was measured (STAI; Spielberger, 1985). Subjects were asked to rate 20 first-person statements describing one's anxiety at this moment from 1='not at all' to 4='very much so'. State anxiety was quantified as a sum across items with higher scores reflecting more anxiety (range=20-80).
Positive-Negative Affect Scale | 1 minute; collected five times throughout each experimental session
  Well-validated measure of self-reported positive and negative affect was measured (PANAS; Watson et al., 1988). Subjects were asked to rate 20 adjectives on a 5-point Likert scale from 1='not at all or very slightly' to 5='extremely'. Two sub-scales were analyzed separately: positive vs. negative affect. Mean scores for each sub-scale were calculated and ranged from 1 to 5 with higher scores reflecting more positive or more negative affect.
Blood pressure | 1 minute; collected six times throughout each experimental session
  Seated and resting systolic and diastolic blood pressure (BP; mmHg) was measured.
Heart Rate | 1 minute; collected six times throughout each experimental session
  Seated and resting heart rate (HR; bpm) was measured.

CONTACTS AND LOCATIONS:
Overall Officials: Eric A Woodcock, PhD, Principal Investigator — Wayne State University
Locations (1):
- Wayne State University, Detroit, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cox LS, Tiffany ST, Christen AG. Evaluation of the brief questionnaire of smoking urges (QSU-brief) in laboratory and clinical settings. Nicotine Tob Res. 2001 Feb;3(1):7-16. doi: 10.1080/14622200020032051. PMID 11260806
- [Background] Spielberger CD. Assessment of state and trait anxiety: Conceptual and methodological issues. Southern Psychologist 2(4): 6-16, 1985.
- [Background] Watson D, Clark LA, Tellegen A. Development and validation of brief measures of positive and negative affect: the PANAS scales. J Pers Soc Psychol. 1988 Jun;54(6):1063-70. doi: 10.1037//0022-3514.54.6.1063. PMID 3397865
- [Background] Hughes JR, Hatsukami D. Signs and symptoms of tobacco withdrawal. Arch Gen Psychiatry. 1986 Mar;43(3):289-94. doi: 10.1001/archpsyc.1986.01800030107013. PMID 3954551